CLINICAL TRIAL: NCT05297916
Title: Early Versus Delayed Postoperative Enteral Feeding to Reduce the Incidence of Perineal Wound Infection Following Anterior Sagittal Anorectoplasty of Congenital Recto-vestibular Fistula
Brief Title: Delayed vs Early Enteral Feeding After Anterior Sagittal Anorectopexy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammad Gharieb Mohammad Khirallah, assistant professor of pediatric surgery, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35054/11/21
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Onset of Perineal Wound Infection
Keywords: recto-vestibular fistula,; early enteral feeding; peripheral parenteral nutrition; perineal wound infection
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: delayed enteral feeding ingroup 1 early enteral feeding in group 2
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- delayed enteral feeding (Active Comparator): delayed enteral feeding
  Interventions: Other: enteral feeding
- early enteral feeding (Active Comparator): early enteral feeding
  Interventions: Other: enteral feeding

INTERVENTIONS:
Other: enteral feeding — to intake oral feeding or delay it

SUMMARY:
to study the effect of early vs delayed enteral feeding following ASARP in females with congenital recto-vestibular fistula

DETAILED DESCRIPTION:
congenital Recto vestibular fistula represents the commonest type of anorectal malformation in females. The treatment of this anomaly is mainly approached either through anterior or posterior sagittal ano-rectoplasty approach. Several perioperative factors may affect the outcome. One of major postoperative complications is the occurrence of wound infection.

Purpose: we aimed to study the effect of delayed vs early postoperative enteral feeding on the occurrence of postoperative wound infection and dehiscence.

Patients and methods:

A prospective randomized trial included 55 infants with recto-vestibular fistula. All infants were managed by single stage anterior sagittal anorectoplasty at an age ≥ 3 months. Patients were divided into two groups. group A included infants who started oral intake on the 5th postoperative day and group B included infants who started oral intake on the 2nd postoperative day. The primary outcome was the onset of perineal wound infection. Group A infants were kept on peripheral parenteral nutrition during fasting period.

ELIGIBILITY:
Inclusion Criteria:

* All female infants with congenital rectoperineal fistula

Exclusion Criteria:

* patients with major anomalies, patients who have staged repair

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-08-02 (Estimated); Study Completion 2022-10-02 (Estimated)

PRIMARY OUTCOMES:
perineal wound infection | WITHIN TWO WEEKS POST OPERATIVE
  the occurrence of wound infection after ASARP

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Egypt